CLINICAL TRIAL: NCT00118339
Title: A Prospective Randomized Pilot Study Using Ice Chips Versus Room Temperature Normal Saline Rinses Orally During Administration of Melphalan to Decrease the Severity and Duration of Oral Mucositis in Patients With Multiple Myeloma Undergoing Autologous Peripheral Blood Stem Cell Transplant
Brief Title: Ice Chips or Saline Mouth Rinse in Reducing or Preventing Mucositis in Patients Receiving Melphalan and Autologous Stem Cell Transplant for Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Purpose: Supportive Care
Other Study IDs: 1845.00; FHCRC-1845.00; CDR0000430699 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2011-09-01 (Estimated); Status verified 2011-08

CONDITIONS: Multiple Myeloma; Plasma Cell Neoplasm
Keywords: oral complications; drug/agent toxicity by tissue/organ; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Drug-Related Side Effects and Adverse Reactions

INTERVENTIONS:
Drug: chemoprotection
Procedure: complementary or alternative medicine procedure
Procedure: management of therapy complications

SUMMARY:
RATIONALE: Chemoprotective agents may protect normal cells from the side effects of chemotherapy. Ice chips or saline mouth rinse may lessen the severity or help prevent symptoms of mucositis or mouth sores in patients receiving melphalan and autologous stem cell transplant for multiple myeloma. It is not yet known whether ice chips are more effective than saline mouth rinse in reducing or preventing mucositis.

PURPOSE: This randomized phase III trial is studying ice chips to see how well they work compared to saline mouth rinse in reducing or preventing mucositis in patients receiving melphalan and autologous stem cell transplant for multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of administering ice chips vs room temperature normal saline oral rinse before, during, and after melphalan administration, in terms of reducing or eliminating grade 3 or 4 oral mucositis, in patients undergoing autologous peripheral blood stem cell transplantation (PBSCT) for multiple myeloma.
* Compare the number of days that IV narcotic therapy is required for oral mucositis pain in patients treated with these regimens.
* Compare the use of IV hydration and/or total parenteral nutrition after autologous PBSCT in patients treated with these regimens.
* Compare overall quality of life, in terms of ability to eat food and drink liquids, in patients treated with these regimens.

OUTLINE: This is a randomized, pilot study. Patients are stratified according to age (less than 60 years vs 60 years and over). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral ice chips 15 minutes before, during, and for 8 hours after melphalan infusion* on day -2.
* Arm II: Patients receive room temperature normal saline oral rinses over 30 seconds 15 minutes before, during, and for 8 hours after melphalan infusion* on day -2.

All patients undergo autologous peripheral blood stem cell transplantation (PBSCT)* on day 0.

NOTE: *Patients receive melphalan infusion and undergo autologous PBSCT on protocol FHCRC-1137.00.

Quality of life is assessed 3 days a week for 4 weeks.

After completion of study treatment, patients are followed for 28 days and then periodically thereafter.

PROJECTED ACCRUAL: A total of 40 patients (20 per treatment arm) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma
* Scheduled to undergo an autologous peripheral blood stem cell transplantation (PBSCT) for multiple myeloma on protocol FHCRC-1137.00

  * Scheduled to receive a regimen of single-agent melphalan at a dose of 200 mg/m^2 before PBSCT

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No concurrent artificial saliva on the day of melphalan infusion (day -2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William I. Bensinger, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States